CLINICAL TRIAL: NCT03380598
Title: An Evaluation of a Web-based CLinical Obesity Support System (CLOSS) - A Randomized Trial of Childhood Obesity Treatment
Brief Title: An Evaluation of a Web-based System for Optimization of Behavioral Childhood Obesity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, PhD Pediatric Nurse, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOSS100
Record Dates: First submitted 2017-11-08; First posted 2017-12-21 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Childhood Obesity
Keywords: Mobile Health, Self-Monitoring, Behavioural Treatment
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care according to regular treatment routines at the clinic during 6 months.
  Interventions: Behavioral: Usual care
- CLOSS (Active Comparator): Usual care plus using a web based support system for self-monitoring weight at physical activity.
  Interventions: Behavioral: CLOSS

INTERVENTIONS:
Behavioral: CLOSS — Usual care plus using mobile application's to register weight and physical activity as well as for communication with the clinic. A web-based system enables health care professionals to follow the the patient's daily weight registration online.
  Arms: CLOSS
Behavioral: Usual care — Usual care. The child and parent(s) at regular visits to the nurse at the clinic
  Arms: Usual care

SUMMARY:
This study evaluates the families' and health care professional's experience from using a web based support system including mobile applications for self-monitoring weight and physical activity. Changes in BMI standard deviation score are compared between usual care (control) and usual care with complementary web-based support system (intervention).

DETAILED DESCRIPTION:
In this study children with obesity were randomized to either usual care according to regular routine (control group) or to usual care plus a web-based support system (intervention group). The system is based on a smartphone application connected to a scale and an activity measuring wrist-band. Data is automatically transferred from the accessories to the smartphone, where data is presented graphically. The data is transferred to the clinic for support. The system is developed for communication between the clinic and family. The randomization was done at the start of individual treatment and lasted for 6 months. Investigators studied the families and health care professional's experience of using the web-based support system as well as changes in BMI standard deviation score in the control and intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Obesity according to International Obesity Task Force (IOTF)
* Swedish speaking parents
* Parents able to use a smart phone
* No pharmacological treatment that could intervene the obesity treatment

Exclusion Criteria:

* Diagnosed with or undergoing assessment of neuropsychiatric disorder
* Structured obesity treatment the past 6 months
* Hypothalamic obesity

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

PRIMARY OUTCOMES:
Familie's experience and feasibility of the treatment | 6 months after baseline
  CLOSS specific questionnaire, control vs intervention

SECONDARY OUTCOMES:
Health care professional's required working time for control vs intervention | During the intervention 6 months
  Time report
Health care professional's experience using the web based support system | During the intervention 3 and 6 months
  CLOSS specific questions regarding the application

OTHER OUTCOMES:
Change in BMI Standard Deviation Score | During the intervention 3 and 6 months
  Control vs intervention
Familie's compliance | During the intervention 6 months
  Control - visits to the clinic Intervention - daily weighing, daily usage of accelerometer, and visits to the clinic

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson, PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - National Childhood Obesity Center, Karolinska University hospital, Huddinge
  - Outpatient paediatric clinic at Norrtälje Hospital, Norrtälje
  - Outpatient paediatric clinic at Södertälje Hospital, Södertälje

REFERENCES:
- [Derived] Johansson L, Hagman E, Danielsson P. A novel interactive mobile health support system for pediatric obesity treatment: a randomized controlled feasibility trial. BMC Pediatr. 2020 Sep 23;20(1):447. doi: 10.1186/s12887-020-02338-9. PMID 32967638